CLINICAL TRIAL: NCT01084941
Title: Lifestyle Intervention to Limit Excessive Weight Gain During Pregnancy in Minority Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guillermo Umpierrez (Other)
Responsible Party: Sponsor-Investigator, Guillermo Umpierrez, Professor of Medicine, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00030742
Record Dates: First submitted 2010-03-09; First posted 2010-03-11 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-07

CONDITIONS: Pregnancy; Weight Gain
Keywords: pregnancy; weight gain; obesity; pregnancy and weight gain
MeSH Terms: conditions — Weight Gain; Obesity; Gestational Weight Gain | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle intervention (Experimental): Women on the intervention group will participate in a lifestyle program based on diet and moderate physical activity implemented shortly after first recognition of pregnancy. These women will attend monthly nutrition and physical activity educational sessions, and receive booster every 2 weeks.
  Interventions: Behavioral: Lifestyle Intervention group
- Standard of care group (Active Comparator): Patients randomized to the standard of care group will receive counseling routinely provided to all prenatal care women as recommended by the Institute of Medicine for appropriate nutrition and weight gain and ACOG guidelines for appropriate physical activity during pregnancy.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Lifestyle Intervention group — Women on the intervention group will participate in a lifestyle program based on diet and moderate physical activity implemented shortly after first recognition of pregnancy. These women will attend monthly nutrition and physical activity educational sessions, and receive booster every 2 weeks.
  Arms: Lifestyle intervention
Behavioral: Standard of Care — Patients randomized to the standard of care group will receive counseling routinely provided to all prenatal care women as recommended by the Institute of Medicine for appropriate nutrition and weight gain and ACOG guidelines for appropriate physical activity during pregnancy.
  Arms: Standard of care group

SUMMARY:
The prevalence of overweight and obesity is increasing among pregnant women in the United States. More than one-third of women of reproductive age in the US are overweight or obese, and two thirds of women gain more weight in pregnancy than is recommended by the Institute of Medicine guidelines. Maternal obesity during pregnancy increases the risk of complications to both mother and child. Minority women (Blacks and Hispanics) have higher rates of overweight and obesity when they become pregnant, experience higher rates of excessive weight gain during pregnancy, and experience higher rates of maternal and neonatal complications after adjusting for sociodemographic characteristics and comorbidities than Caucasian women. Epidemiologic studies indicate that lifestyle modification programs based on diet and exercise are promising approaches in controlling weight gain as well as in preventing type 2 diabetes in populations at risk. We hypothesize that overweight/obese minority women (Blacks and Hispanics) assigned to a culturally-grounded lifestyle intervention program based on diet and moderate exercise will result in higher compliance with Institute of Medicine guidelines for weight gain than women receiving standard care. Such lifestyle modifications should reduce risk of maternal and neonatal complications. We propose 1) to determine whether a lifestyle intervention program, based on diet and moderate physical activity implemented shortly after first recognition of pregnancy, will result in higher compliance with Institute of Medicine guidelines for weight gain compared to women receiving standard care; 2) to determine the occurrence of carbohydrate intolerance and GDM at 24-28 weeks gestation (after the first 10-12 weeks of intervention) and at 6 weeks postpartum between women in the lifestyle intervention group and women receiving standard care; and 3) to explore the impact of the lifestyle intervention on the development of maternal and fetal complications during pregnancy. By limiting excessive weight gain, the lifestyle intervention program may prevent the burden of obesity-related complications during pregnancy and reduce risk of subsequently developing overt diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Blacks and Hispanic
* women between 18-45 years of age;
* 2) overweight and obese (BMI > 25 kg/m2),
* 3) have a sedentary lifestyle (<30 minutes/day of moderate physical activity), and
* 4) prenatal care established at less than 20 weeks of gestation,
* 5) with a singleton pregnancy.

Exclusion Criteria:

* Women with 1) age < 18 or > 45 years,
* 2) > 20 weeks gestation,
* 3) history of diagnosis of type 2 diabetes, hypertension, cardiovascular disease, chronic renal disease, and active liver disease (AST > 3 ULN),
* 4) anemia (hemoglobin < 10 g, hematocrit < 32%);
* 5) current medications which adversely influence glucose tolerance (corticosteroids),
* 6) multiple pregnancy,
* 7) women not planning to continue pregnancy to term, 7) contraindications to participate in regular physical activity,
* 8) patients with mental conditions rendering them unable to understand the nature, scope, and possible consequences of the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2010-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome is whether a woman's weight gain follows the Institute of Medicine's recommendations for pregnancy weight gain. | 36 weeks

SECONDARY OUTCOMES:
To compare the occurrence of carbohydrate intolerance and GDM at 24-28 weeks gestation and after delivery between women in the lifestyle intervention group and women receiving standard care. | 36 weeks
To explore the impact of the lifestyle intervention in preventing maternal and fetal complications between women in the lifestyle intervention group and women receiving standard care. | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States